CLINICAL TRIAL: NCT03334279
Title: Detection of Field Cancerization in the Clinically Normal Oral Mucosa of Cannabis and Cigarette Smokers (Ex-vivo Study)
Brief Title: Effect of Cannabis and Cigarette Smoking on Oral Mucosa
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Abdelwahed Kotb, assistant lecturer, oral and maxillofacial pathology- cairo university, Cairo University
Other Study IDs: CEBD-CU_2017-10-27
Record Dates: First submitted 2017-10-21; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-10

CONDITIONS: Field Cancerization for Cannabis Smokers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- non smokers
- cigarette smokers: Cigarette smokers to be included in the study must be frequent smokers (at least 10 cigarettes a day) for a period not less than 5 years.
  Interventions: Other: Cigarette smokers
- simultaneous cigarette and cannabis smokers: frequent cigarette smokers (at least 10 cigarettes a day) and frequent cannabis smoker (at least 3 times/week) for not less than 5 years.
  Interventions: Other: Simultaneous cigarette and cannabis smokers

INTERVENTIONS:
Other: Cigarette smokers — frequent cigarette smoking for not less than 5 years
  Groups: cigarette smokers
Other: Simultaneous cigarette and cannabis smokers — frequent cigarette and cannabis smoking for not less than 5 years
  Groups: simultaneous cigarette and cannabis smokers

SUMMARY:
The aim of this study is to detect P53 expression in clinically normal oral mucosa of cigarette smokers, simultaneous cigarette and cannabis smokers and non-smokers as a surrogate marker for field cancerization.

DETAILED DESCRIPTION:
Roles and Responsibilities:

1. Ali Abd El Wahed Abd El Fatah Kotb (A.K.) operator, data enterer, Assistant lecturer, Oral and Maxillofacial Pathology, Faculty of Oral and Dental Medicine, Cairo university, Egypt.
2. Professor Dr. Heba Dahmoush (H.D.) main supervisor, data monitoring,auditing professor, Oral and Maxillofacial Pathology, Faculty of Oral and Dental Medicine, Cairo university, Egypt.
3. Eman Desoky (E.D.) sample size calculation, statistician,Faculty of Oral and Dental Medicine, Cairo University, Egypt.
4. Evidence Based Dentistry Committee (CEBD)help in reporting study protocol following SPIRIT guidelines,Faculty of Oral and Dental Medicine, Cairo University, Egypt.
5. Research Ethics Comittee (CREC)protocol reviewer in order to protect the right, safety, dignity and well-being of the participants, Faculty of Oral and Dental Medicine, Cairo University, Egypt.

1- Intervention: A.K. will collect specimens from cigarette smokers and simultaneous cigarette and cannabis smokers. then the expression of p53 as a marker for field cancerization will be investigated in formaline fixed paraffine embedded specimens of mucosal biopsies obtained from the oral mucosa of both groups.

2-comparator: mucosal biopsies from non smokers will be investigated as a copmaratitive to smokers group.

ELIGIBILITY:
Inclusion Criteria:

* frequent smokers (at least 10 cigarettes a day) for a period not less than 5 years.
* Simultaneous smokers to be included in the study must be frequent cigarette smokers (at least 10 cigarettes a day) for a period not less than 5 years plus frequent cannabis smoker (at least 3 times per week) for a period not less than 5 years.

Exclusion Criteria:

* Exposure to other carcinogens.
* un-clear smoking history.
* medically compromised patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: routine patients already coming for simultaneous dental or surgical procedures..
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
P53 expression as a surrogate marker for field cancerization | not less than 5 years
  The areas containing the most uniformly stained tissues will be chosen for evaluation in area-area/area-percent measurments